CLINICAL TRIAL: NCT06600048
Title: Spinal Anesthesia by Hyperbaric Prilocaine in Day-Case Perianal Surgery: A Randomized Controlled Trial
Brief Title: Spinal Anesthesia by Hyperbaric Prilocaine in Day-Case Perianal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSharkawy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264PR839/9/24
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Spinal Anesthesia; Hyperbaric; Prilocaine; Day-Case; Perianal Surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyperbaric prilocaine group (Experimental): Patients will receive 1.5 ml (30 mg) 0.5% hyperbaric prilocaine.
  Interventions: Drug: Hyperbaric prilocaine
- Hyperbaric bupivacaine group (Active Comparator): Patients will receive 1.5 ml (7.5 mg) 0.5% hyperbaric bupivacaine.
  Interventions: Drug: Hyperbaric bupivacaine

INTERVENTIONS:
Drug: Hyperbaric prilocaine — Patients will receive 1.5 ml (30 mg) 0.5% hyperbaric prilocaine.
  Arms: Hyperbaric prilocaine group
Drug: Hyperbaric bupivacaine — Patients will receive 1.5 ml (7.5 mg) 0.5% hyperbaric bupivacaine.
  Arms: Hyperbaric bupivacaine group

SUMMARY:
The aim of this study is to evaluate the effect of spinal anesthesia by hyperbaric prilocaine in day-case perianal surgery.

DETAILED DESCRIPTION:
Day-case spinal anesthesia with short-acting local anesthetics such as lidocaine and chloroprocaine can provide short times to discharge. However, the association of lidocaine with transient neurologic symptoms (TNS) and chloroprocaine with neurologic injury has limited the use of these agents in spinal anesthesia.

Hyperbaric bupivacaine has been used for spinal anesthesia for decades owing to the low incidence of TNS.

Prilocaine is also an amide local anesthetic that has an intermediate duration of action. It is available in the hyperbaric form that can be used for spinal anesthesia in day-case surgeries.

Hyperbaric prilocaine provides faster spinal block onset and earlier patient recovery in ambulatory surgery compared to plain prilocaine.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years.
* Both sexes.
* American Society of Anesthesiology (ASA) physical status I-II.
* Scheduled for perianal surgery under spinal anesthesia.

Exclusion Criteria:

* Allergy to the studied drugs.
* Patients with contraindications to spinal anesthesia.
* Patients with advanced cardiac, renal, or hepatic diseases.
* Previous voiding difficulty.
* Patients taking anticholinergic medications.
* Time of surgery exceeds 75 min.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-09-17 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Time till home readiness | 24 hours postoperatively
  The time-to-home readiness will be assessed as the time from the end of surgery until the patients reached a post-anesthesia discharge score (PADS) ≥9 and were able to void spontaneously or receive a urinary catheter, and the sensory block resolved to the S3 dermatome.

SECONDARY OUTCOMES:
Time to block regression | 6 hours postoperatively
  The time to block regression will be from intrathecal injection until sensation is regained at the S1 dermatome.
Time of onset of motor block | Intraoperatively
  The time of onset of the motor block will be assessed from intrathecal injection of local anesthetic until a grade 3 Bromage score is achieved
Time to spontaneous voiding | 24 hours postoperatively
  Time to spontaneous voiding will be recorded.
Time to the 1st rescue analgesia | 24 hours postoperatively
  Time to the first request for the rescue analgesia will be recorded from end of surgery to first dose of pethidine administrated
Total ketorolac consumption | 24 hours postoperatively
  Total ketorolac consumption will be recorded. If the numerical rating scale (NRS) becomes ≥3, 30 mg ketorolac IM will be given when needed (maximum every six hours).
Heart rate | Every 10 min till the end of surgery (up to 1 hour)
  Heart rate will be recorded throughout the operation: every 5 minutes for the first 15 minutes and every 10 minutes until the end of the surgery.
Mean arterial pressure | Every 10 min till the end of surgery (up to 1 hour)
  Mean arterial pressure will be recorded throughout the operation: every 5 minutes for the first 15 minutes and every 10 minutes until the end of the surgery.
Incidence of adverse events | 24 hours postoperatively
  Incidence of adverse events such as postoperative nausea and vomiting (PONV), voiding difficulty, or any other complication.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.